CLINICAL TRIAL: NCT00695474
Title: Vitamin D and Type 2 Diabetes - a Cross Sectional Study
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Regionshospitalet Silkeborg (Other)
Responsible Party: MD, Med. Sci. Lotte Oerskov, Medical Department, Silkeborg Hospital
Other Study IDs: M-20080061
Record Dates: First submitted 2008-06-09; First posted 2008-06-11 (Estimated); Last update posted 2009-07-14 (Estimated); Status verified 2009-07

CONDITIONS: Hypovitaminosis D; Type 2 Diabetes Mellitus
Keywords: Hypovitaminosis D; Type 2 diabetes; Glycemic control; Inflammation; Blood pressure
MeSH Terms: conditions — Vitamin D Deficiency; Diabetes Mellitus, Type 2; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples, urine.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: The cohort consists of type 2 diabetics from the outpatient clinic at Silkeborg Hospital.

SUMMARY:
The purpose of the study is to describe vitamin D status among patients with type 2 diabetes and to determine the association between serum 25-hydroxyvitamin D and glycemic control, markers of inflammation and blood pressure

DETAILED DESCRIPTION:
It has been estimated that 1 billion people worldwide have vitamin D deficiency or insufficiency. It is well known that vitamin D deficiency causes osteoporosis, increases the risk of fracture and causes muscle weakness. But there is now evidence that calcium malnutrition and hypovitaminosis D are predisposing conditions for various common chronic diseases such as malignancies (particularly colon, breast and prostate) chronic inflammatory and autoimmune disease (inflammatory bowel disease, multiple sclerosis) as well as metabolic disorders (metabolic syndrome, hypertension).

It has also been reported that vitamin D deficiency may predispose to glucose intolerance, altered insulin secretion and type 2 diabetes mellitus.

The purpose of this study is to determine vitamin D status among type 2 diabetics in our outpatient clinic and examine the relationship between vitamin D status , calcium and phosphorous metabolism, inflammatory markers, glycemic control, blood pressure and lipid profile.

Moreover the patients are asked to answer a questionnaire regarding lifestyle, exercise, sun exposure and food intake.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Patients of Danish extraction
* Written consent

Exclusion Criteria:

* Renal failure (Urea > 12 mmol/l)
* Age < 18 years
* malabsorption

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of Danish type 2 diabetics from the outpatient clinic at Silkeborg Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2008-06; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Vitamin D status and its association with inflammation, glycemic control, lipids and blood pressure. | December 08

SECONDARY OUTCOMES:
Lifestyle (exercise, sun exposure, food intake) | December 08

CONTACTS AND LOCATIONS:
Overall Officials: Lotte Oeskov, MD, Principal Investigator — Medical Department, Silkeborg Hospital, Falkevej 1-3, 8600 Silkeborg, Denmark